CLINICAL TRIAL: NCT00995488
Title: ABX209: Phase II Trial of Combination ABI-007, Carboplatin, and Gemcitabine for First Line Treatment of Advanced Urothelial Cancer.
Brief Title: Trial of Combination ABI-007, Carboplatin, and Gemcitabine for First Line Treatment of Advanced Urothelial Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated prematurely due to low accrual.
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009.025; HUM00029138 (Other: University of Michigan Medical IRB (IRBMED))
Record Dates: First submitted 2009-10-14; First posted 2009-10-15 (Estimated); Results first posted 2014-09-19 (Estimated); Last update posted 2015-09-11 (Estimated); Status verified 2015-08

CONDITIONS: Urothelial Cancer; Bladder Cancer
Keywords: Urothelial Cancer; ABI-007; Bladder Cancer; front-line
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ABI-007 (Experimental): ABI-007 combined with Carboplatin, and Gemcitabine
  Interventions: Drug: ABI-007 (Abraxane®)

INTERVENTIONS:
Drug: ABI-007 (Abraxane®) — ABI-007 is a novel albumin-bound paclitaxel combining a protein with a chemotherapeutic agent in the particle form.
  Other Names: Abraxane; albumin-bound paclitaxel

SUMMARY:
This study will evaluate the safety and efficacy of the combination of ABI-007, carboplatin and gemcitabine in the treatment of patients with advanced bladder cancer.

Study participants will have been diagnosed with advanced bladder cancer. Cisplatin based chemotherapy in this setting has activity but is not curative. Furthermore, patients with this disease have comorbidities that limit the use of cisplatin based therapy. Combination paclitaxel, carboplatin and gemcitabine is active and well tolerated in this patient population.

Paclitaxel is formulated with ethanol and a Cremophor EL (polyoxyethylated castor oil) which contribute to the side effects associated with paclitaxel. ABI-007 (brand name Abraxane™) is a form of paclitaxel that does not contain these additives and may deliver more drug to tumor cells. ABI-007 is approved by the United States Food and Drug Administration (FDA) in the treatment of metastatic (advanced) breast cancer based on superior anticancer effect, and is being evaluated in other cancers in research studies.

DETAILED DESCRIPTION:
On the basis of the known single agent activity of paclitaxel in urothelial cancer, the activity of combination therapy with paclitaxel, carboplatin, and gemcitabine in advanced urothelial cancer coupled with the results from studies in breast cancer demonstrating improved clinical efficacy of ABI-007 over paclitaxel with a more favorable toxicity profile, we propose this phase II trial evaluating the efficacy and safety of the combination of ABI-007, carboplatin, and gemcitabine in patients with advanced urothelial cancer.

Carboplatin and gemcitabine dosing and schedule is based on our previous trial of paclitaxel, carboplatin, and gemcitabine which showed acceptable toxicity.

Due to the extent of hematologic toxicities expected with this combination and reported with weekly schedules of ABI-007 based combinations as well as our experience on UMCC protocol 2007.061 which originally utilized a weekly ABI-007 with gemcitabine and carboplatin, we do not feel continuous weekly dosing will be feasible. Therefore this trial is designed with ABI-007 on a D1 only schedule every 21 days. The starting dose of ABI-007 will be 220 mg/m2, because of the risk of significant bone marrow suppression, with the option of a dose escalation in patients who tolerate therapy well after the first cycle to 260 mg/m2 every 21 days.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients at least 18 years of age.
* Histologic or cytologic diagnosis of urothelial carcinoma (transitional cell carcinoma either pure or mixed histology) that is metastatic or locally recurrent or locally advanced and not eligible for higher priority trials.
* must have measurable disease.
* Patients must have recovered from any radiation therapy and must not have had more than 25% of the bone marrow irradiated.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2 (Appendix 1.)
* Life expectancy of at least 12 weeks.
* Adequate organ and marrow function as defined below obtained within 14 days from registration:

  * absolute neutrophil count >1,500/µL
  * platelets >100,000/µL
  * total bilirubin =1.5 mg/dL
  * creatinine <2.0 mg/dL
  * AST and ALT <2.5 X upper limits of normal
* Timing guideline for pre-study labs and measurements:

  * All pre-study labs required for determination of eligibility are to be completed within 14 days prior to registration.
  * X-rays and/or scans to assess all disease sites are to be completed within 1 month prior to registration (or the next business day if falls on a weekend or holiday).
* All patients must be informed of the investigational nature of this study and must sign an informed consent in accordance with institutional and federal guidelines.

Exclusion Criteria:

* Previous systemic chemotherapy for the current stage of disease.
* Prior treatment with ABI-007 or other taxane (prior treatment with taxane in neoadjuvant or adjuvant setting more than one year prior to registration is allowed).
* Pre-existing neuropathy that is > grade 2 (i.e. interfering with patient function).
* History of or known spinal cord compression, or carcinomatous meningitis, or evidence of symptomatic brain or leptomeningeal disease on screening CT or MRI scan.
* Known HIV positive patients may not participate. This is to avoid additional complications that immune suppression and HIV infection may cause due to the intense nature of the chemotherapy in this trial.
* Concurrent treatment on another therapeutic clinical trial. Supportive care trials or non-treatment trials, e.g. QOL, are allowed.
* Pregnancy or breastfeeding. Female subjects must be surgically sterile or be postmenopausal, or must agree to use effective contraception during the period of therapy. All female subjects with reproductive potential must have a negative pregnancy test (serum) prior to enrollment. Male subjects must be surgically sterile or must agree to use effective contraception during the period of therapy. The definition of effective contraception will be based on the judgment of the principal investigator or a designated associate.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the investigator would make the subject inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2009-10; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maha Hussain, MD, Principal Investigator — University of Michigan Medical School/Internal Medicine Dept.
Locations (1):
- University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan, United States

REFERENCES:
- [Result] Alva A, Daignault S, Smith DC, Hussain M. Phase II trial of combination nab-paclitaxel, carboplatin and gemcitabine in first line therapy of advanced urothelial carcinoma. Invest New Drugs. 2014 Feb;32(1):188-94. doi: 10.1007/s10637-013-0054-5. Epub 2013 Dec 10. PMID 24318901

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ABI-007
Started | 16
Completed | 15
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | ABI-007
Number analyzed (Participants) | 16
Age, Continuous [Median (Full Range); unit: years] | 73.9 [51.3 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 13
Histology [Number; unit: participants] — Participant tumor histology at the start of the study.
  participants
    Pure Urothelial | 13
    Mixed Urothelial with Squamous | 2
    Mixed Urothelial with Adenocarcinoma | 1
Primary Site [Number; unit: participants] — The site of cancer origin.
  participants
    Bladder | 13
    Ureter/ Renal Pelvis | 3
Disease Status [Number; unit: participants] — The status of the disease at baseline (locally advanced or metastatic).
  participants
    Metastatic | 13
    Locally Advanced or Recurrent Unresectable | 3
GFR [Number; unit: participants] — GFR at baseline. Glomerular filtration rate (GFR) is a test used to check how well the kidneys are working.
  participants
    Greater than or Equal to 60 mL/min | 9
    Less than 60 mL/min | 7
ECOG Performance Status [Number; unit: participants] — The Eastern Cooperative Oncology Group (ECOG) performance status is the measure of a patients general well being and activities of daily life. The scoring system runs from 0 to 5 where 0 represents perfect health and 5 represents death.
  participants
    0 | 4
    1 | 11
    2 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Partial or Complete Response
Description: Clinical efficacy of ABI-007 based therapy will be determined by the overall response rate (Partial Response [PR] + Complete Response[CR]) to therapy.
  Partial Response: At least a 30% decrease in the sum of the longest diameter (LD) of target lesions.
  Complete Response: Disappearance of all target lesions.
Time Frame: 2 years
Population: 16 participants began treatment however one patient withdrew from the study and was therefore not evaluable.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ABI-007
Number analyzed (Participants) | 15
percentage of participants | 6.3 [0.2 to 32]

2. Secondary Outcome: Median Overall Survival
Description: The Median Overall Survival was captured in months.
Time Frame: 2 years
Population: 16 participants began treatment however one patient withdrew from the study and was therefore not evaluable.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | ABI-007
Number analyzed (Participants) | 15
months | 13.1 [9.8 to 19.6]

ADVERSE EVENTS:
Arm/Group | ABI-007
Serious Adverse Events (participants affected / at risk) | 11/16
Other Adverse Events (participants affected / at risk) | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ABI-007 (N=16)
ADH Secretion Abnormality (SIADH) (Endocrine disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 2 (2)
Cardiac ischemia/infarction : Acute myocardial infarction (Cardiac disorders) | 1 (1)
Congestive Heart Failure (Cardiac disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dissease Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Hemarthrosis (Vascular disorders) | 1 (1)
Hemorrhage:GI (Gastrointestinal disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Hypotension (Cardiac disorders) | 2 (2)
Infection (Infections and infestations) | 1 (1)
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (Infections and infestations) | 1 (1)
Infection documented microbiologically with Gr 3 or 4 neutrophils (Infections and infestations) | 1 (1)
Infection-documented clinically with Gr 4 neutrophils- Skin (cellulitis) (Infections and infestations) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3)
Mucositis (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Pain-Back (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain-Chest wall (Cardiac disorders) | 1 (1)
Photophobia (Eye disorders) | 1 (1)
Syncope (General disorders) | 2 (2)
Ventricular Arrhythmia-Ventricular tachycardia (Cardiac disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
hyponatermia (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ABI-007 (N=16)
ALT Increase (Investigations) | 4 (4)
AST increase (Investigations) | 2 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 9 (10)
Anorexia (Metabolism and nutrition disorders) | 5 (5)
Leukocytopenia (Blood and lymphatic system disorders) | 14 (24)
Anemia (Blood and lymphatic system disorders) | 16 (33)
Lymphopenia (Blood and lymphatic system disorders) | 13 (18)
Nausea (Gastrointestinal disorders) | 6 (8)
Neuropathy:Sensory (Nervous system disorders) | 4 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 16 (38)
constipation (Gastrointestinal disorders) | 4 (4)
creatinine increase (Investigations) | 3 (3)
dizziness (Nervous system disorders) | 2 (2)
fatigue (General disorders) | 12 (17)
hyperglycemia (Metabolism and nutrition disorders) | 7 (8)
hyponatremia (Metabolism and nutrition disorders) | 2 (2)
increase creatinine (Investigations) | 2 (2)
neutropenia (Blood and lymphatic system disorders) | 9 (21)
pain (General disorders) | 2 (2)
vomiting (Gastrointestinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes